CLINICAL TRIAL: NCT07328100
Title: A Randomized, Double-blind, Parallel Controlled Clinical Trial to Evaluate the Efficacy of Coenzyme I for Injection in the Treatment of Vascular Aging（Pilot Stydy）
Brief Title: Efficacy and Safety of Coenzyme I for Injection on Vascular Aging.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Senior doctor, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAD-VA
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Vascular Aging; NAD
MeSH Terms: interventions — NAD; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Drug: Coenzyme I for Injection
- Control Group (Placebo Comparator)
  Interventions: Drug: NaCl (placebo)

INTERVENTIONS:
Drug: Coenzyme I for Injection — Subjects receive 7 consecutive days of intravenous infusion of Coenzyme I for injection.
  Arms: Intervention Group
Drug: NaCl (placebo) — Subjects receive 7 consecutive days of intravenous infusion of NaCl(0.9%).
  Arms: Control Group

SUMMARY:
Emerging evidence identifies vascular aging independently predicting cardiovascular events, yet effective clinical interventions remain lacking. Nicotinamide adenine dinucleotide (NAD+) is an essential cofactor whose levels decline with age, and preclinical studies suggest that boosting NAD+ can improve vascular function and structure. Preliminary clinical studies in healthy older adults indicate that supplementation with NAD+ precursors, such as nicotinamide riboside(NR) or nicotinamide mononucleotide (NMN), can reduce arterial stiffness as measured by pulse wave velocity (PWV). However, whether NAD+ supplementation can improve vascular endothelial function and exert anti-stiffening effects in patients who have already developed measurable arterial stiffness remains unknown. Based on this evidence, the investigator hypothesize that the Coenzyme I for Injection will reverse vascular aging in older adults with established arterial stiffening.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 40-70 years;
2. cf-PWV was abnormally elevated and above the upper limit of its age-and blood-pressure matched reference range;
3. Systolic Blood Pressure < 160 mmHg and ≥ 140 mmHg or Diastolic BP < 100 mmHg ≥ 90mmHg;
4. Signed informed consent.

Exclusion Criteria:

1. Consumption of foods or medications containing high levels of NAD+, NR, NAM, NMN, or niacin-related components (including Vitamin B3 and natural health products) within 3 months prior to screening；
2. History of major cardiovascular or cerebrovascular events, including myocardial infarction, angina, stroke, or hospitalization for arterial revascularization；
3. Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg；
4. Diagnosis of malignant tumor；
5. Known allergy or history of severe adverse reactions to Coenzyme I injection or any of its components；
6. History of severe allergies or infusion reactions；
7. Women who are pregnant, breastfeeding, or planning pregnancy；
8. Severe hepatic or renal dysfunction: ALT or AST > 5 times the upper limit of normal; glomerular filtration rate ≤ 30 mL/min/1.73 m²；
9. Concurrent participation in another clinical trial without completion of the follow-up period；
10. Other conditions deemed by the investigator as unsuitable for inclusion, such as psychiatric or psychological disorders.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in flow-mediated vasodilation(FMD) | Day 8/28
  Changes in FMD from baseline to day 8/28.

SECONDARY OUTCOMES:
Changes in cf-PWV. | day 8/28
  Changes in cf-PWV from baseline to day 8/28.
Changes in retinal arteriovenous ratio (AVR) and wall/lumen ratio (WLR) | day 8/28
  Changes in retinal arteriovenous ratio (AVR) and wall/lumen ratio (WLR) from baseline to day 8/28.
Changes in the level of NAD+ | day 8/28
  Changes in the level of NAD+ from baseline to day 8/28.
Changes in the metabolomics. | day 8/28
  Changes in the metabolomics from baseline to day 8/28.
Changes in office blood pressure and 24-hour ambulatory blood pressure | day 8/28
  Changes in office blood pressure and 24-hour ambulatory blood pressure from baseline to day 8/28.
The change in the urine albumin-to-creatinine ratio | day 8/28
  The change in the urine albumin-to-creatinine ratio from baseline to day 8/28.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China